CLINICAL TRIAL: NCT04196933
Title: Temporal Synthesis of Vestibular and Extra-Vestibular Sensory Signals
Brief Title: Analysis of Vestibular Compensation Following Clinical Intervention for Vestibular Schwannoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Following further collection and analysis of temporal binding data, we found the relationship between PSS and clinical outcomes to not be strong enough for adaptation.
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Oregon Health and Science University (Other); University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Richard Lewis, Associate Professor, Otolaryngology and Neurology; Director, Jenks Vestibular Laboratory, Massachusetts Eye and Ear Infirmary
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2018P003117; 1R01DC017425-01 (NIH)
Record Dates: First submitted 2019-12-06; First posted 2019-12-12 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-06

CONDITIONS: Migraine; Vestibular Migraine; Vestibular Schwannoma; Motion Sickness; Dizziness; Vestibular Disorder
Keywords: sensory integration; cochlear implant; vestibular implant; balance; dizziness; vestibular disorders
MeSH Terms: conditions — Migraine Disorders; Neuroma, Acoustic; Motion Sickness; Dizziness; Vestibular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Normal Controls (No Intervention): normal control subjects - no history of neurologic or inner ear disease
  The investigators will characterize vestibular spatial and temporal precision by calculating perceptual thresholds for vestibular (yaw rotation) stimuli in normal subjects over a wide age range. Vestibular-visual temporal binding is then performed on each subject and the relationship between the principal parameters (vestibular perceptual thresholds [inversely related to spatial precision] and the PSS and TBW from the temporal binding paradigm) will be examined. The investigators will collect qualitative assessments of dizziness/disbalance (DHI: dizziness handicap index) and quantitative measurements of balance and vestibular function (FGA: functional gait analysis, postural sway, and standard rotational testing - VOR gain, time constant, asymmetry).
- Central Vestibular Dysfunction (No Intervention): Migraine and Vestibular Migraine patients
  The investigators intend to evaluate vestibular (yaw rotation) - visual temporal binding in people with a wide range of motion sickness sensitivities (as quantified with standard questionnaires), including normal subjects, people with migraine and with vestibular migraine.
- Peripheral Vestibular Dysfunction (No Intervention): Vestibular Schwannoma patients
  The basic approach is to characterize the precision of their vestibular information (i.e., perceptual thresholds for spatial precision), and their temporal binding characteristics for vestibular (yaw rotation)-visual inputs, in three states: pre-op, sub-acute post-op (2-6 weeks), and chronic post-op (6 months+). At each state the investigators will also assess the quality of their vestibular-mediated behaviors through questionnaires (e.g. DHI), postural sway, functional gait analysis, and standard rotational testing (VOR gain, time constant, and asymmetry).
- Implant Subjects (Experimental): Cochlear Implant (CI)/Vestibular Implant (VI) patients
  A causative role for vestibular precision in temporal binding will be investigated in the VI patients, since the noise characteristics of the vestibular channel will be varied and to determine how this affects thresholds and temporal binding. As part of a second aim, the investigators will use VI and CI prosthetic signals in patients who have never received them together to see how the brain process sensory cues to which it is essentially naïve. Finally, after the acute experiments the investigators will provide 8 hours of 'physiologic' VI and CI stimulation by turning both implants on, sound modulates activity in the CI as usual, and angular head motion modulates activity in the VI while the subject actively explores the hospital environment.
  Interventions: Behavioral: Temporal Binding Adaptation - PSS adaptation with VI stimulation; Behavioral: Chronic Motion-modulated Stimulation
- Post-op Vestibular Schwannoma patients (Experimental): Vestibular Schwannoma patients who are 6mos+ post-surgery (for removal of vestibular schwannoma, resulting in 8th nerve being cut & complete loss of peripheral vestibular signals from affected ear). While many post-op VS patients recover well, some continue to have persistent problems with balance and symptoms of dizziness. This study will explore how/whether PSS adaptation may improve vestibular clinical outcomes such as improved gait and dizziness symptoms following gait with horizontal (yaw) head motion.
  Interventions: Behavioral: Temporal Binding Adaptation - PSS training

INTERVENTIONS:
Behavioral: Temporal Binding Adaptation - PSS training — After the PSS and TBW are calculated with the standard TOJ paradigm, 100 training trials are provided where the SOA is set to a PSS slightly greater than what was the mean calculated for normal subjects, with the goal of shifting the PSS in a direction associated with better clinical vestibular parameters and vestibular precision measurements (e.g. standard rotational testing VOR time constant, lower DHI, higher FGA score) . Then the TOJ task will be repeated but every 10 testing trials will be followed by 10 training trials (SOA = PSS desired or mean normal PSS), and this pattern will be repeated 10 times to 100 more training trials interspersed with the Post TOJ data. Subjects will respond after all trials and testing and training will not be distinguished. After this is completed, the new PSS and TBW are calculated. Sham PSS training will be identical to the above except that the 'training' period will consist of random SOAs rather than a series of fixed SOAs.
  Arms: Post-op Vestibular Schwannoma patients
Behavioral: Temporal Binding Adaptation - PSS adaptation with VI stimulation — The adaptation will utilize the same approach used in non-implanted patients. The investigators will provide a repeated, fixed SOA with either the CI or VI leading the other stimulus by 220 ms. After the training period, which will match the number of stimuli pairs provided to our normal vestibular-auditory control subjects undergoing PSS adaptation, the TOJ study is repeated to recalculate the PSS and TBW.
  Arms: Implant Subjects
Behavioral: Chronic Motion-modulated Stimulation — To provide 8 hours of 'physiologic' CI and VI inputs during normal activities, the investigators will employ standard motion-modulated stimulation with the VI. This requires pre-adaptation to a 200 pps tonic stimulation rate (to emulate the push-pull design of the native vestibular system allowing modulating stimulation upward or downward with opposite directions of motion). The three electrodes are connected to the head-mounted prosthetic circuit, which consists of three angular velocity sensors (one aligned with the sensitive axis of each canal) such that head rotations in the plane of the given canal modulate the stimulation rate of the corresponding electrode, upward (for ipsi) or downward (for contralateral) head rotations, thereby simulating normal canal-mediated modulations.
  Arms: Implant Subjects

SUMMARY:
Multiple sensory cues are typically generated by discrete events, and while they do not reach the cerebrum simultaneously, the brain can bind them temporally if they are interpreted as corresponding to a single event. The temporal binding of vestibular and non-vestibular sensory cues is poorly understood and has not been studied in detail, despite the fact that the vestibular system operates in an inherently multimodal environment. In this study, the researchers are investigating the physiology and pathophysiology of vestibular temporal binding by studying normal subjects, patients with peripheral and central vestibular dysfunction, and patients with vestibular and cochlear signals provided by prosthetic implants in the inner ear.

DETAILED DESCRIPTION:
Multiple sensory cues are generated by discrete events (e.g., the vestibular-visual signals after hitting a pothole) and while they do not reach the cerebrum simultaneously, the brain can synthesize them if they are interpreted as corresponding to a single event. This is critical because the central representation of an event is improved if two or more relevant cues are integrated but conversely is degraded if unrelated inputs are synthesized. Little research has focused on temporal binding of vestibular signals with other sensory cues, even though the vestibular system operates in an inherently multimodal environment, and virtually nothing is known about temporal binding abnormalities in patients with peripheral or central vestibular disorders. The investigators will use psychophysical tests (quantifying the PSS [point of subjective simultaneity] and TBW [temporal binding window]) to study vestibular temporal binding in normal people, patients with combined vestibular and cochlear prostheses, and patients with peripheral or central vestibular dysfunction. The researchers will investigate two fundamental aspects of temporal binding: its dependence on signal precision and adaptation driven by habitual exposure to sensory patterns. Furthermore, the researchers will investigate how and why temporal binding differs from normal in patients with peripheral and central vestibular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Normal subjects

* normal vestibular-oculomotor exams
* normal low-frequency standard rotational testing
* normal hearing

Migraine

* meets International Headache Society (IHS) criteria for migraine with or without aura
* tested more than 2 weeks after most recent migraine headache

Vestibular Migraine

* meets Barany Society criteria for vestibular migraine, which includes:
* episodic vestibular symptoms that occur with headaches that meet the IHS criteria for migraine
* tested more than 2 weeks after most recent migraine headache or vestibular episode

Vestibular Schwannoma

* existence of unilateral vestibular schwannoma (pre & post clinical intervention e.g. surgical resection)
* must plan to have clinical intervention such as sub-occipital surgical approach with complete sectioning of the vestibular nerve
* rotational testing to assess pre-surgical vestibular function
* audiogram
* brain MRI consistent with vestibular schwannoma
* audiography in each ear

Vestibular (VI) and Cochlear (CI) Implant subjects

* scheduled for CI surgery because of deafness
* minimum 5 year history of documented absence of auditory and vestibular function, based on review of their audiograms and vestibular tests
* specific vestibular criteria: peak ice water caloric response of less than 3deg/s for each ear; yaw VOR time constant <3s and gain <0.25; and reduced head impulse gain (<0.25) for all canal planes
* specific audiographic criteria: 80dB or greater sensorineural hearing loss in both ears

Exclusion Criteria:

Normal subjects

* history of otologic or neurologic disease
* on vestibular suppressant medication (benzodiazepine, antihistamine, anticholinergic)
* pregnant or recently (<6mos) pregnant

Migraine

* history of vestibular symptoms (other than motion sickness)
* evidence of other neurologic or otologic dysfunction
* on migraine prophylactic medications
* on vestibular suppressant medication (benzodiazepine, antihistamine, anticholinergic)

Vestibular Migraine (VM)

* other neurologic or otologic dysfunction as defined above except for central eye movement findings that are consistent with VM and therefore not exclusionary.
* on migraine prophylactic medication
* on vestibular suppressant medication (benzodiazepine, antihistamine, anticholinergic)

Vestibular Schwannoma

* other otologic disease (other than presbycusis) or any neurologic disease (other than migraine)
* on vestibular suppressant medication (benzodiazepine, antihistamine, anticholinergic)

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in postural sway/balance | baseline and post-PSS adaptation (1 hour)
  Measurements of postural sway during Romberg testing on floor and foam (including an extra 60s balance test during which subject stands on foam and shakes head left and right at 1hz frequency while fixating on a point a set distance away) pre & post temporal binding adaptation (TBW & PSS training).
Change in rapid measure of gait | baseline and post-PSS adaptation (1 hour)
  This measure is scored before and after PSS adaptation in UVD (unilateral vestibular dysfunction) patients. Gait is scored by performance on a task derived from the FGA (walking 40 feet while turning the head from side to side). It is scored on a 0 to 10 visual scale and provides a rapid assessment of vestibular function pre and post adaptation.
Change in measure of inducible dizziness | baseline and post-PSS adaptation (1 hour)
  Looking at the change between before and after PSS adaptation in UVD (unilateral vestibular dysfunction) patients. Inducible dizziness is the symptom severity provoked by a task derived from the FGA (walking 40 feet while turning the head from side to side). It is scored on a 0 to 10 visual scale and provides a rapid assessment of vestibular function pre and post adaptation.
Change in Point of Subjective Simultaneity (PSS) | baseline and 1 hour post 8-hour VI-CI 'physiologic' stimulation
  Pre and post chronic motion-modulated stimulation in CI/VI patients - the PSS will be measured during temporal binding testing

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States